CLINICAL TRIAL: NCT01541826
Title: The Effect of Chokeberry Polyphenols on Biomarkers of Cardiovascular Disease and Antioxidant Defenses in Former Smokers
Brief Title: Study of Chokeberry to Reduce Cardiovascular Disease Risk in Former Smokers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Connecticut (Other)
Responsible Party: Principal Investigator, Bradley Bolling, Assistant Professor, University of Connecticut
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: H11-311; 120068 (Other: University of Connecticut)
Record Dates: First submitted 2012-02-24; First posted 2012-03-01 (Estimated); Results first posted 2017-07-11 (Actual); Last update posted 2017-07-11 (Actual); Status verified 2017-04

CONDITIONS: Cardiovascular Disease; Oxidative Stress
Keywords: aronia; LDL cholesterol; polyphenols; bioavailability; oxidative stress
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Color-matched rice powder pill (Placebo Comparator): Color-matched rice powder pill
  Interventions: Dietary Supplement: Placebo capsule
- Chokeberry extract capsule (Active Comparator): Chokeberry extract capsule
  Interventions: Dietary Supplement: Chokeberry Extract
- Chokeberry extract capsule (acute) (Experimental): Chokeberry extract capsule pharmacokinetics
  Interventions: Dietary Supplement: Chokeberry extract capsule, acute

INTERVENTIONS:
Dietary Supplement: Chokeberry Extract — Consumption of 2 x 250 mg chokeberry extract capsules daily for 12 weeks.
  Arms: Chokeberry extract capsule
Dietary Supplement: Placebo capsule — Color-matched rice powder pill, 2 x 250 mg/day for 12 weeks
  Arms: Color-matched rice powder pill
Dietary Supplement: Chokeberry extract capsule, acute — Chokeberry extract capsule, 2 x 250 mg, one-time dose.
  Arms: Chokeberry extract capsule (acute)

SUMMARY:
The purpose of this project is to determine whether chokeberry polyphenols mitigate cardiovascular disease risk in former smokers.

DETAILED DESCRIPTION:
More than 31% of Connecticut adults are former smokers, which may contribute to the high cardiovascular disease (CVD) risk in this state. Atherosclerosis, a hallmark of CVD, is a progressive life-long process. Chronic cigarette smoking increases atherosclerosis and CVD risk. While smoking cessation may lower CVD risk, former smokers still are at high CVD risk. The mechanisms by which smoking accelerates atherosclerosis formation are not fully understood. This knowledge gap prevents development of informed interventions to reduce CVD risk in former smokers.

Previous work suggests smoking increases oxidative stress and leads to elevated CVD risk. Former smokers also have decreased antioxidants and markers of vascular function in the circulation, suggesting that despite cessation, smoking has a lingering adverse effect on CVD protective mechanisms. Chokeberry (Aronia melanocarpa) is a native Connecticut plant rich in polyphenol antioxidants and is a promising intervention for reducing CVD risk in former smokers. Chokeberries have diverse polyphenols such as anthocyanins, proanthocyanidins, resveratrol, quercetin, and chlorogenic acid. Chokeberry consumption improves dyslipidemia, inhibits inflammation, and reduces oxidative stress in humans and animals, all of which could contribute to the prevention of CVD in former smokers. Therefore, our central hypothesis is that dietary chokeberry polyphenols reduce CVD risk in former smokers by improving lipid profiles and inhibiting inflammation and oxidative stress. Our long-term goal is to define the mechanisms by which polyphenol antioxidants mitigate CVD risk. The overall goal of this project is to conduct a randomized placebo-controlled clinical trial to evaluate the cardio-protective effects of dietary chokeberry polyphenols in former smokers.

Our objectives are to determine 1) the effect of chokeberry polyphenols on plasma cholesterol and triglyceride levels and on gene expression involved in cholesterol metabolism; 2) the extent to which chokeberry improves antioxidant and vascular function in former smokers; and 3) the association of bioavailability of chokeberry polyphenols to changes in biomarkers of CVD risk.

Successful completion of this work will result in improved understanding of the role of dietary berry polyphenols to regulate lipid metabolism, inflammation and oxidative stress. Thus, this study will be an important step to developing dietary recommendations for individuals predisposed to CVD risk, particularly former smokers.

ELIGIBILITY:
Inclusion Criteria:

* Former smoker (previously smoked ≥3 cigarettes/day for at least 1 year, cessation for at least 6 months
* Healthy male or female between 18-65 y
* Serum clinical ranges no more than mildly elevated (serum cholesterol <240 mg/dL) and serum triglyceride (<150 mg/dL)
* Resting blood pressure <140/90 mm Hg
* Stable body weight (±5 lb) for last 2 months
* BMI ranges within normal and overweight (18.5-39 kg/m2)
* Willing to maintain normal exercise level (<7 h/wk)
* Willing to avoid exercise 24 h prior to blood sampling
* Willing to ingest a dietary chokeberry supplement or placebo (500 mg/d) daily for 12 wks.

Exclusion Criteria:

* Previous diagnoses of CVD, diabetes, or arthritis (except for osteo-arthritis)
* Currently being treated for cancer (i.e., chemotherapy, radiation therapy)
* Women with prescribed estrogen replacement therapy
* Practicing slimming diet
* Practicing vegetarian diet
* Currently taking vitamin or mineral supplements or plant pills
* Alcohol consumption exceeding the definition of moderate drinking (2 drinks/day or a total of 12/week for men or 1 drink/day or a total of 7/week for women)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2012-02; Primary Completion 2015-08 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bradley W Bolling, PhD, Principal Investigator — University of Connecticut, University of Wisconsin-Madison
Locations (1):
- Roy E. Jones Building, Storrs, Connecticut, United States

REFERENCES:
- [Result] Xie L, Lee SG, Vance TM, Wang Y, Kim B, Lee JY, Chun OK, Bolling BW. Bioavailability of anthocyanins and colonic polyphenol metabolites following consumption of aronia berry extract. Food Chem. 2016 Nov 15;211:860-8. doi: 10.1016/j.foodchem.2016.05.122. Epub 2016 May 19. PMID 27283706
- [Result] Xie L, Vance T, Kim B, Lee SG, Caceres C, Wang Y, Hubert PA, Lee JY, Chun OK, Bolling BW. Aronia berry polyphenol consumption reduces plasma total and low-density lipoprotein cholesterol in former smokers without lowering biomarkers of inflammation and oxidative stress: a randomized controlled trial. Nutr Res. 2017 Jan;37:67-77. doi: 10.1016/j.nutres.2016.12.007. Epub 2016 Dec 10. PMID 28215316

RESULTS

PARTICIPANT FLOW:
Groups:
- Chokeberry Extract Capsule: Chokeberry extract capsule
  Chokeberry Extract: Consumption of 2 x 250 mg chokeberry extract capsules daily for 12 weeks.
  Chokeberry extract capsule, acute: Chokeberry extract capsule, 2 x 250 mg, one-time dose.
- Chaokeberry Extract Capsule (Acute): Chokeberry extract capsule, acute: Chokeberry extract capsule, 2 x 250 mg, one-time dose.
Period: Overall Study
Arm/Group | Color-matched Rice Powder Pill | Chokeberry Extract Capsule | Chaokeberry Extract Capsule (Acute)
Started | 28 | 28 | 6
Completed | 24 | 25 | 6
Not Completed | 4 | 3 | 0
Not completed — Lost to Follow-up | 2 | 3 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Color-matched Rice Powder Pill | Chokeberry Extract Capsule | Chokeberry Extract Capsule (Acute) | Total
Number analyzed (Participants) | 24 | 25 | 6 | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.4 (14.8) | 32.6 (12.7) | 31.3 (12.8) | 34.9 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 12 | 3 | 28
  Male | 11 | 13 | 3 | 27
Height [Mean (Standard Deviation); unit: m] | 1.73 (0.92) | 1.71 (0.83) | 1.74 (0.97) | 1.72 (0.87)
Average years of smoking [Mean (Standard Deviation); unit: years] — Population: Missing value for one participant in acute study.
  years
    number analyzed (Participants) | 24 | 25 | 5 | 54
    (all) | 14.9 (11.9) | 8.96 (6.68) | 4.8 (3.0) | 11.9 (10.0)
Degree of past smoking [Count of Participants; unit: Participants] — Population: Missing value for one participant in acute study.
  Participants
    3-5 cigarettes/day: number analyzed (Participants) | 24 | 25 | 5 | 54
    3-5 cigarettes/day | 2 | 4 | 1 | 7
    6-10 cigarettes/day: number analyzed (Participants) | 24 | 25 | 5 | 54
    6-10 cigarettes/day | 4 | 7 | 1 | 12
    11-15 cigarettes/day: number analyzed (Participants) | 24 | 25 | 5 | 54
    11-15 cigarettes/day | 4 | 4 | 2 | 10
    16-20 cigarettes/day: number analyzed (Participants) | 24 | 25 | 5 | 54
    16-20 cigarettes/day | 11 | 6 | 0 | 17
    >20 cigarettes/day: number analyzed (Participants) | 24 | 25 | 5 | 54
    >20 cigarettes/day | 3 | 4 | 1 | 8
Weight [Mean (Standard Deviation); unit: kg] | 81.5 (17.2) | 77.2 (21.1) | 72.8 (9.5) | 79.3 (19.2)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 27.2 (4.7) | 25.7 (5.0) | 24.1 (2.3) | 26.5 (4.9)
Waist circumference [Mean (Standard Deviation); unit: cm] | 86.0 (17.1) | 90.9 (35.1) | 79.4 (8.4) | 88.5 (27.6)
Systolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 121 (14) | 117 (16) | 111.3 (7.7) | 119 (15)
Diastolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 76.0 (10.4) | 75.3 (12.0) | 73.3 (4.7) | 75.6 (11.0)
Total cholesterol [Mean (Standard Deviation); unit: mg/dL] | 203 (36) | 220 (63) | 160 (30) | 213 (51)
HDL-cholesterol [Mean (Standard Deviation); unit: mg/dL] | 28.7 (6.1) | 26.8 (7.6) | 54.8 (15.7) | 27.6 (6.9)
LDL-cholesterol [Mean (Standard Deviation); unit: mg/dL] | 158 (30) | 175 (54) | 99.2 (19.2) | 168 (44)
Triglycerides [Mean (Standard Deviation); unit: mg/dL] | 82.1 (37.3) | 89.6 (45.4) | 69.2 (27.1) | 86.3 (41.0)
Total cholesterol/HDL cholesterol [Mean (Standard Deviation); unit: dimensionless ratio] | 7.3 (1.5) | 8.5 (2.7) | 3.2 (0.7) | 8.0 (2.3)

OUTCOME MEASURES:

1. Primary Outcome: LDL Cholesterol
Description: Change in LDL cholesterol from baseline after chronic supplementation. Not determined in Chokeberry Extract Capsule (Acute) arm as this arm was a one-time dose.
Time Frame: Baseline, 6 weeks, 12 weeks of intervention
Population: Not determined in Chokeberry Extract Capsule (Acute) arm as this arm was a one-time dose.
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Color-matched Rice Powder Pill | Chokeberry Extract Capsule
Number analyzed (Participants) | 24 | 25
mg/dL
  6 weeks | 0.9 (4.2) | -12.6 (5.3)
  12 weeks | -0.4 (5.9) | -18.5 (7.8)

2. Secondary Outcome: Total Cholesterol
Description: Change in fasting total cholesterol from baseline after chronic supplementation. Not determined in Chokeberry Extract Capsule (Acute) arm as this arm was a one-time dose.
Time Frame: 6 and 12 weeks after supplementation
Population: Not determined in Chokeberry Extract Capsule (Acute) arm as this arm was a one-time dose.
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Color-matched Rice Powder Pill | Chokeberry Extract Capsule
Number analyzed (Participants) | 24 | 25
mg/dL
  Baseline | 203 (7) | 220 (13)
  6 weeks (change from baseline) | -0.1 (4.6) | 1.4 (2.5)
  12 weeks (change from baseline) | -1.3 (6.4) | -17.9 (7.6)

3. Secondary Outcome: HDL-cholesterol
Description: Change in fasting plasma cholesterol from baseline after chronic supplemenation. Not determined in Chokeberry Extract Capsule (Acute) arm as this arm was a one-time dose.
Time Frame: 6 and 12 weeks after supplementation
Population: Not determined in Chokeberry Extract Capsule (Acute) arm as this arm was a one-time dose.
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Color-matched Rice Powder Pill | Chokeberry Extract Capsule
Number analyzed (Participants) | 24 | 25
mg/dL
  Baseline | 28.8 (1.3) | 26.8 (1.5)
  6 weeks (change from baseline) | -0.9 (1.0) | 0.2 (0.8)
  12 weeks (change from baseline) | -0.7 (1.4) | 0.2 (0.8)

4. Secondary Outcome: Triglycerides
Description: Change in fasting plasma triglycerides from baseline after chronic supplementation. Not determined in Chokeberry Extract Capsule (Acute) arm as this arm was a one-time dose.
Time Frame: 6 and 12 weeks after supplementation
Population: Not determined in Chokeberry Extract Capsule (Acute) arm as this arm was a one-time dose.
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Color-matched Rice Powder Pill | Chokeberry Extract Capsule
Number analyzed (Participants) | 24 | 25
mg/dL
  Baseline | 82.1 (7.6) | 89.6 (9.0)
  6 weeks (change from baseline) | -0.6 (2.7) | 1.0 (5.9)
  12 weeks (change from baseline) | -1.0 (5.9) | 2.0 (8.5)

5. Secondary Outcome: Resting Systolic Blood Pressure
Description: Change in resting systolic blood pressure after chronic supplementation. Not determined in Chokeberry Extract Capsule (Acute) arm as this arm was a one-time dose.
Time Frame: Baseline, 6 weeks, and 12 weeks following intervention
Population: Not determined in Chokeberry Extract Capsule (Acute) arm as this arm was a one-time dose.
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Color-matched Rice Powder Pill | Chokeberry Extract Capsule
Number analyzed (Participants) | 24 | 25
mmHg
  Baseline | 121 (3) | 117 (3)
  6 weeks (change from baseline) | -0.8 (1.5) | 2.8 (1.7)
  12 weeks (change from baseline) | 0.2 (2.9) | 1.2 (2.4)

6. Secondary Outcome: Resting Diastolic Blood Pressure
Description: Change in resting diastolic blood pressure after chronic supplementation. Not determined in Chokeberry Extract Capsule (Acute) arm as this arm was a one-time dose.
Time Frame: Baseline, 6 weeks, and 12 weeks following intervention
Population: Not determined in Chokeberry Extract Capsule (Acute) arm as this arm was a one-time dose.
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Color-matched Rice Powder Pill | Chokeberry Extract Capsule
Number analyzed (Participants) | 24 | 25
mmHg
  Baseline | 76.0 (2.1) | 75.3 (2.4)
  6 weeks (change from baseline) | -1.2 (2.4) | 5.0 (1.3)
  12 weeks (change from baseline) | -1.1 (1.7) | 2.0 (1.5)

7. Secondary Outcome: Urinary F2-isoprostanes
Description: Change in resting urinary F2-isoprostanes after chronic supplementation. Not determined in Chokeberry Extract Capsule (Acute) arm as this arm was a one-time dose.
Time Frame: Baseline and 12 weeks following intervention
Population: Not determined in Chokeberry Extract Capsule (Acute) arm as this arm was a one-time dose.
Measure: Mean (Standard Error); unit: ng/mmol creatinine
Arm/Group | Color-matched Rice Powder Pill | Chokeberry Extract Capsule
Number analyzed (Participants) | 24 | 25
ng/mmol creatinine
  Baseline | 71.0 (8.1) | 58.6 (7.0)
  12 weeks | 81.6 (7.8) | 68.4 (9.0)

8. Secondary Outcome: 3-hydroxy-3-methyl-glutaryl Coenzyme A Reductase (HMGR)
Description: Monocyte messenger ribonucleic acid (mRNA) expression normalized to glyceraldehyde-3-phosphate dehydrogenase (GAPDH) after chronic supplementation. Not determined in Chokeberry Extract Capsule (Acute) arm as this arm was a one-time dose.
Time Frame: Baseline, 12 wk
Population: Not determined in Chokeberry Extract Capsule (Acute) arm as this arm was a one-time dose.
Measure: Mean (Standard Error); unit: relative expression (HMGR/GAPDH)
Arm/Group | Color-matched Rice Powder Pill | Chokeberry Extract Capsule
Number analyzed (Participants) | 24 | 25
relative expression (HMGR/GAPDH)
  Baseline | 0.90 (0.06) | 0.91 (0.06)
  12 weeks | 1.16 (0.28) | 0.79 (0.12)

9. Secondary Outcome: LDL Receptor (LDLR)
Description: Monocyte LDL receptor mRNA normalized to glyceraldehyde-3-phosphate dehydrogenase after chronic supplementation. Not determined in Chokeberry Extract Capsule (Acute) arm as this arm was a one-time dose.
Time Frame: Change from baseline at 12 weeks
Population: Not determined in Chokeberry Extract Capsule (Acute) arm as this arm was a one-time dose.
Measure: Mean (Standard Error); unit: relative expression (LDLR/GAPDH)
Arm/Group | Color-matched Rice Powder Pill | Chokeberry Extract Capsule
Number analyzed (Participants) | 24 | 25
relative expression (LDLR/GAPDH)
  Baseline | 0.90 (0.07) | 0.84 (0.07)
  12 weeks | 0.93 (0.22) | 0.88 (0.26)

10. Secondary Outcome: LDL Receptor (LDLR) Protein
Description: Monocyte LDL receptor protein by Western blot, normalized to β-actin after chronic supplementation. Not determined in Chokeberry Extract Capsule (Acute) arm as this arm was a one-time dose.
Time Frame: Baseline, 12 weeks
Population: Not determined in Chokeberry Extract Capsule (Acute) arm as this arm was a one-time dose.
Measure: Mean (Standard Error); unit: relative expression (LDLR/β-actin)
Arm/Group | Color-matched Rice Powder Pill | Chokeberry Extract Capsule
Number analyzed (Participants) | 24 | 25
relative expression (LDLR/β-actin)
  Baseline | 1.71 (0.33) | 1.45 (0.06)
  12 weeks | 2.47 (0.80) | 1.45 (0.64)

11. Secondary Outcome: Plasma Area Under the Curve of Chokeberry Polyphenols and Their Metabolites.
Description: Plasma area under the curve of chokeberry polyphenols and their metabolites. Measurement (time 0) began at study baseline. Not determined in chronic arms (Color-matched Rice Powder Pill or Chokeberry Extract Capsule).
Time Frame: 0, 0.5, 1, 2, 4, 6, 9, 12, and 24 hours following dose
Population: Not determined in chronic arms (Color-matched Rice Powder Pill or Chokeberry Extract Capsule) as this analysis required additional collection time-points that were not utilized in the other arms.
Measure: Mean (Standard Error); unit: micrograms x h/mL
Arm/Group | Chokeberry Extract Capsule (Acute)
Number analyzed (Participants) | 6
micrograms x h/mL
  Protocatechuic acid | 0.054 (0.013)
  Hippuric acid | 22.350 (4.441)
  3-(4-Hydroxyphenyl)propionic acid | 2.725 (2.391)
  Cyanidin-3-O-glucoside | 0.462 (0.170)
  Peonidin-3-O-galactoside | 0.627 (0.198)

12. Secondary Outcome: Urinary Excretion of Polyphenols
Description: Urinary excretion of polyphenols, from 0 to 24 h after consumption of extract, area under the curve (AUC) in Chokeberry Extract Capsule (acute) arm only.
Time Frame: 0 to 24 h after consumption of extract
Population: as for outcome 11
Measure: Mean (Standard Error); unit: mg x h/mg creatinine
Arm/Group | Chokeberry Extract Capsule (Acute)
Number analyzed (Participants) | 6
mg x h/mg creatinine
  Protocatechuic acid | 3.682 (0.587)
  3,4-dihyrdoxyphenylacetic acid | 11.426 (0.881)
  Hippuric acid | 2429.852 (360.197)
  3-(4-hydroxyphenyl)propionic acid | 2.299 (0.715)
  Cyanidin-3-O-galactoside | 0.016 (0.005)
  Cyanidin-3-O-glucoside | 0.118 (0.070)
  Cyanidin-3-O-arabinoside | 0.088 (0.031)
  Peonidin-3-O-galactoside | 0.053 (0.012)

13. Secondary Outcome: Adiponectin
Description: Fasting plasma adiponectin after chronic consumption. Not determined in Chokeberry Extract Capsule (Acute) arm as this arm was a one-time dose.
Time Frame: Baseline, 6 weeks, 12 weeks
Population: Not determined in Chokeberry Extract Capsule (Acute) arm as this arm was a one-time dose.
Measure: Mean (Standard Error); unit: micrograms/mL
Arm/Group | Color-matched Rice Powder Pill | Chokeberry Extract Capsule
Number analyzed (Participants) | 24 | 25
micrograms/mL
  Baseline | 13.2 (1.9) | 12.8 (1.5)
  6 weeks | 14.2 (2.0) | 13.8 (1.7)
  12 weeks | 12.5 (1.6) | 13.2 (1.5)

14. Secondary Outcome: Interleukin-1 Beta
Description: Fasting plasma interleukin-1 beta after chronic consumption. Not determined in Chokeberry Extract Capsule (Acute) arm as this arm was a one-time dose.
Time Frame: Baseline, 6 weeks, 12 weeks
Population: Not determined in Chokeberry Extract Capsule (Acute) arm as this arm was a one-time dose.
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Color-matched Rice Powder Pill | Chokeberry Extract Capsule
Number analyzed (Participants) | 24 | 25
pg/mL
  Baseline | 9.3 (2.4) | 16.2 (8.6)
  6 weeks | 9.5 (2.7) | 17.0 (9.7)
  12 weeks | 10.1 (3.0) | 14.7 (7.4)

15. Secondary Outcome: Interleukin-6
Description: Fasting plasma interleukin-6 after chronic supplementation. Not determined in Chokeberry Extract Capsule (Acute) arm as this arm was a one-time dose.
Time Frame: Baseline, 6 weeks, 12 weeks
Population: Not determined in Chokeberry Extract Capsule (Acute) arm as this arm was a one-time dose.
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Color-matched Rice Powder Pill | Chokeberry Extract Capsule
Number analyzed (Participants) | 24 | 25
pg/mL
  Baseline | 1.94 (0.34) | 4.68 (1.34)
  6 weeks | 1.87 (0.38) | 5.16 (1.54)
  12 weeks | 1.76 (0.29) | 5.34 (1.52)

16. Secondary Outcome: Monocyte Chemoattractant Protein-1
Description: Fasting plasma monocyte chemoattractant protein-1 after chronic supplementation. Not determined in Chokeberry Extract Capsule (Acute) arm as this arm was a one-time dose.
Time Frame: Baseline, 6 weeks, 12 weeks
Population: Not determined in Chokeberry Extract Capsule (Acute) arm as this arm was a one-time dose.
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Color-matched Rice Powder Pill | Chokeberry Extract Capsule
Number analyzed (Participants) | 24 | 25
pg/mL
  Baseline | 97 (6) | 133 (31)
  6 weeks | 96 (5) | 167 (43)
  12 weeks | 91 (5) | 141 (27)

17. Secondary Outcome: Tumor Necrosis Factor-alpha
Description: Fasting plasma Tumor necrosis factor-alpha after chronic supplementation. Not determined in Chokeberry Extract Capsule (Acute) arm as this arm was a one-time dose.
Time Frame: Baseline, 6 weeks, 12 weeks
Population: Not determined in Chokeberry Extract Capsule (Acute) arm as this arm was a one-time dose.
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Color-matched Rice Powder Pill | Chokeberry Extract Capsule
Number analyzed (Participants) | 24 | 25
pg/mL
  Baseline | 4.36 (1.83) | 5.90 (1.63)
  6 weeks | 4.70 (1.89) | 6.44 (1.83)
  12 weeks | 4.86 (1.85) | 6.10 (1.72)

18. Secondary Outcome: C-reactive Protein
Description: Fasting plasma C-reactive protein after chronic supplementation. Not determined in Chokeberry Extract Capsule (Acute) arm as this arm was a one-time dose.
Time Frame: Baseline, 6 weeks, 12 weeks
Population: Not determined in Chokeberry Extract Capsule (Acute) arm as this arm was a one-time dose.
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Color-matched Rice Powder Pill | Chokeberry Extract Capsule
Number analyzed (Participants) | 24 | 25
pg/mL
  Baseline | 2.54 (0.60) | 2.01 (0.34)
  6 weeks | 2.18 (0.42) | 2.32 (0.39)
  12 weeks | 2.24 (0.38) | 2.29 (0.49)

19. Secondary Outcome: Intercellular Adhesion Molecule 1
Description: Fasting plasma intercellular adhesion molecule 1 after chronic supplementation. Not determined in Chokeberry Extract Capsule (Acute) arm as this arm was a one-time dose.
Time Frame: Baseline, 6 weeks, 12 weeks
Population: Not determined in Chokeberry Extract Capsule (Acute) arm as this arm was a one-time dose.
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | Color-matched Rice Powder Pill | Chokeberry Extract Capsule
Number analyzed (Participants) | 24 | 25
ng/mL
  Baseline | 97.1 (7.2) | 96.6 (5.4)
  6 weeks | 97.6 (7.2) | 99.4 (5.7)
  12 weeks | 100 (8) | 97.5 (5.8)

20. Secondary Outcome: Soluble Vascular Cell Adhesion Molecule 1
Description: Fasting plasma soluble vascular cell adhesion molecule 1 after chronic consumption. Not determined in Chokeberry Extract Capsule (Acute) arm as this arm was a one-time dose.
Time Frame: Baseline, 6 weeks, 12 weeks
Population: Not determined in Chokeberry Extract Capsule (Acute) arm as this arm was a one-time dose.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Color-matched Rice Powder Pill | Chokeberry Extract Capsule
Number analyzed (Participants) | 24 | 25
ng/mL
  Baseline | 585 (23) | 601 (31)
  6 weeks | 604 (23) | 622 (31)
  12 weeks | 604 (26) | 599 (27)

21. Secondary Outcome: P-selectin
Description: Fasting plasma P-selectin after chronic supplementation. Not determined in Chokeberry Extract Capsule (Acute) arm as this arm was a one-time dose.
Time Frame: Baseline, 6 weeks, 12 weeks
Population: Not determined in Chokeberry Extract Capsule (Acute) arm as this arm was a one-time dose.
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | Color-matched Rice Powder Pill | Chokeberry Extract Capsule
Number analyzed (Participants) | 24 | 25
ng/mL
  Baseline | 130 (13) | 124 (12)
  6 weeks | 111 (11) | 127 (12)
  12 weeks | 131 (11) | 145 (17)

22. Secondary Outcome: Total Antioxidant Capacity
Description: Fasting plasma total antioxidant capacity after chronic supplementation. Not determined in Chokeberry Extract Capsule (Acute) arm as this arm was a one-time dose.
Time Frame: Baseline, 6 weeks, 12 weeks
Population: Not determined in Chokeberry Extract Capsule (Acute) arm as this arm was a one-time dose.
Measure: Mean (Standard Error); unit: micrograms vitamin C equivalents/mL
Arm/Group | Color-matched Rice Powder Pill | Chokeberry Extract Capsule
Number analyzed (Participants) | 24 | 25
micrograms vitamin C equivalents/mL
  Baseline | 210 (4) | 208 (3)
  6 weeks | 214 (3) | 211 (3)
  12 weeks | 209 (4) | 207 (4)

23. Secondary Outcome: Catalase Activity
Description: Catalase activity after chronic supplementation. Not determined in Chokeberry Extract Capsule (Acute) arm as this arm was a one-time dose.
Time Frame: Baseline, 6 weeks, 12 weeks
Population: Not determined in Chokeberry Extract Capsule (Acute) arm as this arm was a one-time dose.
Measure: Mean (Standard Error); unit: nmol/min/mL
Arm/Group | Color-matched Rice Powder Pill | Chokeberry Extract Capsule
Number analyzed (Participants) | 24 | 25
nmol/min/mL
  Baseline | 41.7 (1.4) | 41.1 (2.1)
  6 weeks | 35.5 (1.2) | 38.7 (1.5)
  12 weeks | 41.7 (2.3) | 41.2 (1.8)

24. Secondary Outcome: Glutathione Peroxidase Activity
Description: Fasting plasma glutathione peroxidase activity after chronic supplementation. Not determined in Chokeberry Extract Capsule (Acute) arm as this arm was a one-time dose.
Time Frame: Baseline, 6 weeks, 12 weeks
Population: Not determined in Chokeberry Extract Capsule (Acute) arm as this arm was a one-time dose.
Measure: Mean (Standard Error); unit: nmol/min/mL
Arm/Group | Color-matched Rice Powder Pill | Chokeberry Extract Capsule
Number analyzed (Participants) | 24 | 25
nmol/min/mL
  Baseline | 2550 (140) | 2550 (140)
  6 weeks | 2560 (130) | 2500 (160)
  12 weeks | 2470 (110) | 2650 (190)

25. Secondary Outcome: Superoxide Dismutase Activity
Description: Fasting plasma superoxide dismutase after chronic supplementation. Not determined in Chokeberry Extract Capsule (Acute) arm as this arm was a one-time dose.
Time Frame: Baseline, 6 weeks, 12 weeks
Population: Not determined in Chokeberry Extract Capsule (Acute) arm as this arm was a one-time dose.
Measure: Mean (Standard Error); unit: units/mL
Arm/Group | Color-matched Rice Powder Pill | Chokeberry Extract Capsule
Number analyzed (Participants) | 24 | 25
units/mL
  Baseline | 1190 (50) | 1180 (40)
  6 weeks | 1190 (50) | 1160 (40)
  12 weeks | 1160 (60) | 1160 (40)

26. Secondary Outcome: Urinary Polyphenol Excretion
Description: Overnight urinary polyphenol excretion after chronic supplementation. Not determined in Chokeberry Extract Capsule (Acute) arm as this arm was a one-time dose.
Time Frame: 12 weeks
Population: Not determined in Chokeberry Extract Capsule (Acute) arm as this arm was a one-time dose.
Measure: Median (Inter-Quartile Range); unit: mg/mg creatinine
Arm/Group | Color-matched Rice Powder Pill | Chokeberry Extract Capsule
Number analyzed (Participants) | 24 | 25
mg/mg creatinine
  Protocatechuic acid | 1.38 [0.94 to 2.08] | 1.20 [0.64 to 2.03]
  3,4-dihydroxyphenylacetic acid | 5.04 [2.36 to 7.45] | 4.56 [2.18 to 9.09]
  Hippuric acid | 133 [104 to 234] | 138 [62 to 292]
  Ferulic acid | 0.68 [0.24 to 1.20] | 0.71 [0.23 to 3.57]
  3-(4-hydroxyphenyl)propionic acid | 3.91 [0 to 9.95] | 3.36 [0 to 9.68]
  Cyanidin-3-O-glucoside | 0 [0 to 0.055] | 0.00907 [0 to 0.1993]
  Cyanidin-3-O-galactoside | 0 [0 to 0.014] | 0.00466 [0 to 0.0341]
  Cyanidin-3-O-arabinoside | 0 [0 to 0.011] | 0 [0 to 0.053]
  Peonidin-3-O-galactoside | 0 [0 to 0] | 0.008 [0 to 0.0106]
  Sum anthocyanins | 0.014 [0 to 0.091] | 0.134 [0.028 to 0.442]

27. Secondary Outcome: Energy-adjusted Nutrient Intake: Carbohydrate, Protein, Fat, Fiber
Description: Energy-adjusted intake based on 3-day dietary recalls, determined by the average of baseline and 12 weeks. Not determined in Chokeberry Extract Capsule (Acute) arm as this arm was a one-time dose.
Time Frame: Baseline, 12 weeks
Population: Survey data were not available for two participants in the "Color-matched rice powder pill" group. Not determined in Chokeberry Extract Capsule (Acute) arm as this arm was a one-time dose.
Measure: Mean (Standard Error); unit: g/day
Arm/Group | Color-matched Rice Powder Pill | Chokeberry Extract Capsule
Number analyzed (Participants) | 22 | 25
g/day
  Carbohydrate | 238 (9) | 241 (9)
  Protein | 89.2 (3.3) | 90.3 (3.1)
  Fat | 27.8 (4.0) | 77.6 (29.5)
  Fiber | 23.5 (1.6) | 21.0 (1.5)

28. Secondary Outcome: Energy Intake
Description: Energy intake reported from 3-day dietary recalls at baseline and 12 weeks, determined by the average of baseline and 12 weeks. Not determined in Chokeberry Extract Capsule (Acute) arm as this arm was a one-time dose.
Time Frame: Baseline, 12 weeks
Population: as for outcome 27
Measure: Mean (Standard Error); unit: kcal/d
Arm/Group | Color-matched Rice Powder Pill | Chokeberry Extract Capsule
Number analyzed (Participants) | 22 | 25
kcal/d | 2230 (735) | 1950 (530)

29. Secondary Outcome: Energy-adjusted Micronutrient Intake
Description: Energy-adjusted micronutrient intake from 3-day dietary recalls at baseline and 12 weeks. Values reported as the average of baseline and 12 weeks. Not determined in Chokeberry Extract Capsule (Acute) arm as this arm was a one-time dose.
Time Frame: Baseline, 12 weeks
Population: as for outcome 27
Measure: Mean (Standard Error); unit: mg/day
Arm/Group | Color-matched Rice Powder Pill | Chokeberry Extract Capsule
Number analyzed (Participants) | 22 | 25
mg/day
  Sodium | 3490 (160) | 3480 (150)
  Calcium | 947 (58) | 1070 (50)
  Iron | 16.9 (1.3) | 16.9 (1.2)
  Vitamin D | 5.0 (0.9) | 7.1 (0.8)
  Vitamin C | 80.9 (12.9) | 90.9 (12.1)
  Vitamin E | 10.6 (1.1) | 10.8 (1.1)

30. Secondary Outcome: Polyphenol Intake
Description: Energy-adjusted polyphenol intake assessed by 3-day dietary recalls at baseline and 12 weeks, values determined by average of baseline and 12 weeks. Not determined in Chokeberry Extract Capsule (Acute) arm as this arm was a one-time dose.
Time Frame: Baseline, 12 weeks
Population: as for outcome 27
Measure: Mean (Standard Error); unit: mg/day
Arm/Group | Color-matched Rice Powder Pill | Chokeberry Extract Capsule
Number analyzed (Participants) | 22 | 25
mg/day
  Isoflavones | 3.9 (2.7) | 8.5 (2.6)
  Flavanols | 73.9 (20.0) | 81.7 (18.7)
  Flavones | 54.1 (29.1) | 50.3 (27.2)
  Flavanones | 28.8 (11.4) | 22.4 (10.7)
  Flavan-3-ols | 20.6 (7.4) | 26.0 (6.9)
  Anthocyanins | 18.2 (5.2) | 26.6 (4.8)
  Proanthocyanidins | 222 (162) | 418 (150)

31. Secondary Outcome: Intake of Dietary Antioxidant Capacity
Description: Energy-adjusted intake of dietary antioxidant capacity determined by 3-day dietary recalls at baseline and 12 weeks. Values reported as average of baseline and 12 weeks. Not determined in Chokeberry Extract Capsule (Acute) arm as this arm was a one-time dose.
Time Frame: Baseline, 12 weeks
Population: as for outcome 27
Measure: Mean (Standard Error); unit: Vitamin C equivalents
Arm/Group | Color-matched Rice Powder Pill | Chokeberry Extract Capsule
Number analyzed (Participants) | 22 | 24
Vitamin C equivalents | 417 (95) | 292 (89)

32. Secondary Outcome: Energy-adjusted Vitamin A Intake
Description: Energy-adjusted vitamin A intake from 3-day dietary recalls at baseline and 12 weeks. Values reported as the average of baseline and 12 weeks. Not determined in Chokeberry Extract Capsule (Acute) arm as this arm was a one-time dose.
Time Frame: Baseline, 12 weeks
Population: as for outcome 27
Measure: Mean (Standard Error); unit: retinol equivalent mcg/day
Arm/Group | Color-matched Rice Powder Pill | Chokeberry Extract Capsule
Number analyzed (Participants) | 22 | 25
retinol equivalent mcg/day | 3280 (740) | 2690 (690)

ADVERSE EVENTS:
Time Frame: During study intervention stage: 16 weeks
Arm/Group | Color-matched Rice Powder Pill | Chokeberry Extract Capsule | Chokeberry Extract Capsule (Acute)
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/28 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/28 | 0/6
Other Adverse Events (participants affected / at risk) | 0/28 | 0/28 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No